CLINICAL TRIAL: NCT00616096
Title: Study of Immunoadsorption to Treat Severe Atopical Dermatitis Associated With Excessively High Serum IgE Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Detlef Zillikens, M. D., Department of Dermatology, University of Lübeck, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAAD01; AZ07-111
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Dermatitis, Atopic
Keywords: Serum Immunoglobulin E above 5000 kU/l
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: immunoadsorption

INTERVENTIONS:
Procedure: immunoadsorption — First cycle: week 1, day 1-5
  Second cycle: week 5, day 1-5

SUMMARY:
The purpose of this study is to determine whether immunoadsorption is effective in the treatment of severe atopic dermatitis associated with excessively high serum IgE levels.

ELIGIBILITY:
Inclusion Criteria:

* Atopical dermatitis
* Total serum IgE level above 5000 kU/l
* IGA score of 3 or above
* No sufficient response to topical corticosteroids/calcineurin inhibitors, UV therapy (at least 4 weeks of therapy), systemic corticosteroids and cyclosporin A (at least 8 weeks of therapy) or no possibility of a prolonged use of this therapy due to adverse events/contraindications
* 18 years of age or above
* Effective contraception during therapy
* Informed consent

Exclusion Criteria:

* Unfavorable conditions for peripheral venous access
* Known hypersensitivity or allergy towards materials used in the adsorber columns
* Adequate anticoagulation not possible (e.g. multiple allergies towards various anticoagulants)
* Extreme bleeding tendency during anticoagulation
* Hypercoagulability
* Severe cardiovascular disease forbidding extracorporeal circulation
* Severe systemic infection
* Serum IgG level below 250 mg/dl
* Severe immunodeficiency (e.g. AIDS)
* Treatment with an ACE inhibitor (discontinue drug at least 72 h before treatment)
* Pregnancy
* Lactation
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism or mental dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evidence of clinical improvement of skin condition, pruritus and sleep disturbance. | 13 weeks

SECONDARY OUTCOMES:
Evidence of reduction of concomitant topical and/or systemic medication. | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Zillikens, M. D., Study Chair — Department of Dermatology, University of Lübeck, Germany
Locations (1):
- Department of Dermatology, University of Lübeck, Lübeck, Schleswig-Holstein, Germany